CLINICAL TRIAL: NCT03778905
Title: The Correlation Between the Length of Stay in Post Acute Care(PAC) and General Improvements in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Willy Chou, Director of physical medicine and rehabiliation, Chi Mei Medical Hospital
Other Study IDs: CMMC10711-J02
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke patient with complete post-acute care hospitalization: This study aims on stroke patients with complete rehabilitative program in post acute care institution and we try to assess their functional improvements after rehabilitative training.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The stroke patients who admitted to post acute care(PAC) institution would undergo regular rehabilitation.

SUMMARY:
Post-Acute Care(PAC) had been inaugurated in Taiwan for almost four years and current essays revealed positive effects upon general improvements in stroke patient after PAC training. During acute phase, a stroke patient would admit to internal medicine or surgical ward and transferred to rehabilitative ward for more intensive therapeutic programs, restoring muscle power and promoting activity of daily life(ADL) ability. Under relative stable condition, the patient would transfer to PAC institution or hospitals afterwards for continuing rehabilitative program if the patient is acknowledged to have rehabilitative potentials. However, there's still lacking of investigation upon whether the length of stay in PAC correlates to general improvements. Thus, stroke patients' functional ability, such as activities of daily living (ADL) function, swallowing ability and so on, as well as their corresponding scales were assessed on the first and last day during PAC hospitalization. Statistical analysis was conducted via SPSS ver21.0 to compare the relationship of improvements in functional ability and the length of stay in PAC. We're looking forward to the final results!

DETAILED DESCRIPTION:
Functional ability in stroke patients are evaluated by following measurements. Activity of daily life (ADL) function was estimated through modified Rankin scale(MRS) and Barthel index(BI), swallowing ability by functional oral intake scale, nutritional status via mini nutritional assessment, life quality through EuroQoL-5D, instrumental ADL function by Lawton-Brody IADL Scale(IADL), balance/coordination via Berg Balance Test, walking speed through Usual Gait Speed, cardiopulmonary capability by Six-Minute Walk Test, occupational mobility (amount use/quality) via Motor Activity Log, language through concise Chinese aphasia test, motor function of upper extremities by Fugl-Meyer Assessment and so on.

ELIGIBILITY:
Inclusion Criteria:

* >18 y/o
* acute onset of stroke within 30 days
* Modified Rankin Scale 2~4

Exclusion Criteria:

* patients refused to join post acute care(PAC) program
* hemodynamic unstable
* disease progression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stroke patient who meet up criteria of >18 y/o, acute onset of stroke within 30 days and Modified Rankin Scale 2~4 as well as complete post acute care(PAC) rehabilitative program.
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-06-22 (Actual)

PRIMARY OUTCOMES:
Activity of daily life function | 35 days
  Activity of daily life function is evaluated by both Barthel index(Range: 0~100 score; higher score indicates better function) and Modified Rankin Scale(Grade 1~6; the lower grade indicates better function). Task-oriented activity of daily life is assessed by Industrial activity of daily life(Range: Male 0~5 score and female 0~8 score; Higher score indicates better function)
Nutritional status | 35 days
  Nutritional status is evaluated by Mini nutritional assessment(Range: 0.0~30.0). Higher score indicates better function
Oral intake function | 35 days
  Oral intake is evaluated by Functional oral intake scale(Range: level 1~7). Higher level indicates better function.
Cardiopulmonary capacity | 35 days
  Cardiopulmonary capacity is evaluated by 6-minute walk test, which requires the patients to walk as much as they can within 6 minutes. Walking length is presented in meters. Longer distance and more meters indicate better function.
Walking speed | 35 days
  Walking speed is evaluated by Usual Gait Speed, which require the patients to walk certain distance and record the time that needed to finish the whole course. Time is presented with seconds. The shorter time and lower seconds indicate better function.
Upper motor hand function | 35 days
  Upper motor hand function is evaluated by Fugl-Meyer assessment(Range 0~44 scores) Higher scores indicate better function.
Life quality | 35 days
  Life quality is evaluated by EuroQoL-5D(Range: 5~15 scores). Lower scores indicate better life quality.
Balance and coordination | 35 days
  Balance and coordination is evaluated by Berg-Balance test(Range: 0~56). Higher scores indicate better function.
Cognition | 35 days
  Cognition is evaluated by Mini-Mental Sate Examination(Range: 0~30 score). Higher scores indicate better cognition.
Speech function | 35 days
  Speech function is evaluated by Concise Chinese Aphasia Test(Range: 1~12 scores). Higher scores indicate better speech function

CONTACTS AND LOCATIONS:
Overall Officials: Willy Chou, MD, MS, Study Director — Chi Mei Medical Hospital
Locations (1):
- Chi Mei Medical Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.